

# CLINICAL STUDY PROTOCOL

CLBS16 (formerly CLBS14)

#### PHASE 2

An Open-Label Exploratory Clinical Study to Evaluate the Safety and Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Artery Disease

PROTOCOL NUMBER: CLBS16-P01 (formerly CLBS14-P01)

ClinicalTrials.gov Identifier: NCT03508609

Version Number: 7

Version Date: 26 August 2019

Study Caladrius Biosciences

Sponsor(s): 110 Allen Road, Second Floor

Basking Ridge, NJ 07920

#### CONFIDENTIALITY STATEMENT

This document is a confidential communication of Caladrius Biosciences, Inc. Receipt of this document constitutes agreement by the recipient that no unpublished information contained herein shall be published or disclosed without prior written approval, except that this document may be disclosed to the appropriate Ethics Committee under the condition that they keep it confidential.

# PROTOCOL APPROVAL FORM

# CLINICAL STUDY PROTOCOL

#### CLBS16-P01

An Open-Label Exploratory Clinical Study to Evaluate the Safety and Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Artery Disease

ClinicalTrials.gov Identifier: NCT03508609

Version Number: 7

Version Date: 26 August 2019



#### 1. PERSONNEL AND FACILITIES



Note: Changes to Personnel and Facilities do not constitute an amendment and will be updated as needed.

## 2. STUDY SYNOPSIS

| Product Name(s) of Active Granulocyte-Colony Stimulating Factor (G-CSF) mobilized peripheral blood derived autologous CD34+ cells CLINICAL CONDITION(S)/INDICATION(S) • Coronary Microvascular Dysfunction PROTOCOL ID CLBS16-P01 PROTOCOL TITLE An Open-Label Exploratory Clinical Study to Evaluate the Safety and Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease | Name of Investigatio | onal CLBS16 |
|---|---|---|
| Ingredient(s) peripheral blood derived autologous CD34+ cells CLINICAL CONDITION(S)/INDICATION(S) Coronary Microvascular Dysfunction PROTOCOL ID CLBS16-P01 PROTOCOL TITLE An Open-Label Exploratory Clinical Study to Evaluate the Safety a Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease Short Title Exploratory study of CLBS16 for Coronary Microvascular Dysfunct STUDY PHASE 2 STUDY OBJECTIVES AND PURPOSE Study Purpose To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | | |
| CLINICAL CONDITION(S)/INDICATION(S) Coronary Microvascular Dysfunction PROTOCOL ID CLBS16-P01 An Open-Label Exploratory Clinical Study to Evaluate the Safety a Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease Short Title Exploratory study of CLBS16 for Coronary Microvascular Dysfunct STUDY PHASE 2 STUDY OBJECTIVES AND PURPOSE Study Purpose To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | Name(s) of Active | Granulocyte-Colony Stimulating Factor (G-CSF) mobilized |
| Coronary Microvascular Dysfunction PROTOCOL ID CLBS16-P01 An Open-Label Exploratory Clinical Study to Evaluate the Safety and Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease Short Title Exploratory study of CLBS16 for Coronary Microvascular Dysfunct STUDY PHASE 2 STUDY OBJECTIVES AND PURPOSE Study Purpose To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | Ingredient(s) | peripheral blood derived autologous CD34+ cells |
| PROTOCOL ID CLBS16-P01 An Open-Label Exploratory Clinical Study to Evaluate the Safety a Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease Short Title Exploratory study of CLBS16 for Coronary Microvascular Dysfunct STUDY PHASE 2 STUDY OBJECTIVES AND PURPOSE Study Purpose To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | CLINICAL CONDITIO | N(S)/INDICATION(S) |
| PROTOCOL TITLE An Open-Label Exploratory Clinical Study to Evaluate the Safety an Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease Short Title Exploratory study of CLBS16 for Coronary Microvascular Dysfunct STUDY PHASE 2 STUDY OBJECTIVES AND PURPOSE Study Purpose • To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective • To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: • Coronary microvascular function as measured by coronary flow reserve | <ul> <li>Coronary Microva</li> </ul> | ascular Dysfunction |
| Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Arter Disease Short Title Exploratory study of CLBS16 for Coronary Microvascular Dysfunct STUDY PHASE 2 STUDY OBJECTIVES AND PURPOSE Study Purpose • To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective • To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: • Coronary microvascular function as measured by coronary flow reserve | PROTOCOL ID | CLBS16-P01 |
| STUDY PHASE STUDY OBJECTIVES AND PURPOSE Study Purpose • To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective • To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: • Coronary microvascular function as measured by coronary flow reserve | PROTOCOL TITLE | Microvascular Dysfunction and Without Obstructive Coronary Artery |
| STUDY OBJECTIVES AND PURPOSE Study Purpose • To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective • To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: • Coronary microvascular function as measured by coronary flow reserve | Short Title | Exploratory study of CLBS16 for Coronary Microvascular Dysfunction |
| To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | STUDY PHASE | 2 |
| To evaluate the bioactivity of intracoronary delivery of autologous CD34+ cells (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | STUDY OBJECTIVES | AND PURPOSE |
| (CLBS16) in patients with coronary microvascular dysfunction (CMD) and without obstructive coronary artery disease, Primary Objective To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease. Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: Coronary microvascular function as measured by coronary flow reserve | Study Purpose | |
| Secondary Objective(s) To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: • Coronary microvascular function as measured by coronary flow reserve | To evaluate the s | |
| To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters: • Coronary microvascular function as measured by coronary flow reserve | | |
| Coronary microvascular function as measured by coronary flow reserve | | |
| Peripheral arterial tonometry (PAT) | parameters: | |
| Peripheral arterial tonometry (PAT) | | |
| | <ul> <li>Peripheral arteria</li> </ul> | al tonometry (PAT) |
| | ! | |
| * | | |
| | | · |

| Study Type | Interventional |
|---|---|
| Control Type | None |
| Study<br>Classification | Safety/Efficacy |
| Blinding<br>Schema | Open-label |
| Study Design | This is a phase 2 open-label clinical study to evaluate the safety, tolerability, and potential bioactivity of CLBS16 in patients with coronary microvascular dysfunction and without obstructive coronary artery disease. Screening Phase Patients who provide informed consent will be screened for eligibility within 60 days before beginning the study treatment phase. Patients mus be on stable medical therapy for 30 days prior to screening and until treatment with CLBS16. |
| | Treatment Phase |
| | Treatment Filase |







Subject currently uses coumadin, plans to use one of these agents during the time frame of the trial 11. Subject tests positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C Subject has active inflammatory disease or autoimmune disease, or is in a chronic immunosuppressive state 13. Recent history of abuse or current abuser of recreational drugs 14. Subject is pregnant or lactating Malignant neoplasm within 5 years prior to screening Subject has participated in another clinical study within 90 days History of sickle cell disease STATISTICAL ELEMENTS Power Estimate This is an exploratory study to estimate the effect of CLBS16 treatment in this population of patients. The main efficacy endpoint of the change in coronary flow reserve (CFR) from baseline to 6 months after treatment will be measured to estimate the efficacy of treatment. Planned Statistical Analysis The primary measurements of CFR will be used to estimate the efficacy of treatment and the overall analysis framework will be paired t tests using baseline (screening value) and 6-month visit data.



#### 3. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| ACE | Angiotensin converting enzyme |
| ACT | Active clotting time |
| AE | Adverse events |
| AESI | Adverse event of special interest |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AMI | Acute myocardial infarction |
| AP | Anterior-posterior |
| APTT | Activated partial thromboplastin time |
| APV | Average peak velocity |
| ASA | Acetyl salicylic acid (aspirin) |
| AST | Aspartate aminotransferase |
| ВМІ | Body mass index |
| BUN | Blood urea nitrogen |
| BW | Body weight |
| CABG | Coronary artery bypass grafting |
| CAD | Coronary artery disease |
| CBC | Complete blood count |
| СС | Cubic centimeter |
| CCS | Canadian Cardiovascular Society |
| CFR | Coronary flow reserve |
| CFR | Code of federal regulations |
| CK | Creatine kinase |
| CLBS16 | Autologous CD34+ cells |
| CMD | Coronary microvascular dysfunction |
| cMRI | Cardiac magnetic resonance imaging |
| CMV-IgM | Cytomegalovirus immunoglobin M |
| CRP | C-reactive protein |
| CRT | Coronary reactivity testing |
| DCM | Dilated cardiomyopathy |
| ECG | Electrocardiography |
| EDMF | Endothelial-dependent microvascular function |
| e-GFR | Estimated glomerular filtration rate |
| EIMF | Endothelial-independent microvascular function |
| EPC | Endothelial progenitor cells |
| FDA | Food and Drug Administration |
| FS | Fractional shortening |

| Abbreviation | Definition |
|--------------------|-----------------------------------------------------|
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte-Colony Stimulating Factor |
| GFR | Glomerular filtration rate |
| HBc antibody | Hepatitis C surface antigen |
| HBs antigen | Hepatitis B surface antigen |
| hCG | Human chorionic gonadotrophin |
| HCV | Hepatitis C virus |
| HDL | High-density lipoprotein |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human immunodeficiency virus |
| hsCRP | High sensitivity C-reactive protein |
| HTLV-1 | Human T-lymphotrophic virus-1 |
| ICH | International Council on Harmonisation |
| IHD | Ischemic heart disease |
| INR | International normalized ratio |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| IRT | Interactive Response Technologies |
| ITT | Intent-to-treat |
| KDR | Kinase insert Domain Receptor |
| LAD | Left anterior descending |
| LDH | Lactate dehydrogenase |
| LDL | Low-density lipoprotein |
| LpPLa2 | Lipoprotein-associated phospholipase A2 |
| LV | Left ventricular |
| LVEF | Left ventricular ejection fraction |
| MESA | Multi-Ethnic Study of Atherosclerosis |
| mKCCQ | Modified Kansas City Cardiomyopathy Questionnaire |
| MNC | Mononuclear cells |
| NTG | Nitroglycerin |
| NT-proBNP | N-terminal pro B-type natriuretic peptide |
| Parvovirus B19-IgM | Parvovirus B19-IgM |
| PAT | Peripheral arterial tonometry |
| PCI | Percutaneous coronary intervention |
| PET | Positron emission tomography |
| PT | Prothrombin time |

| Abbreviation | Definition |
|---|---|
| QWISE | Study of Quinapril in Women with Chest Pain, Coronary Flow Reserve<br>Limitations and Evidence of Myocardial Ischemia |
| RAO | Right anterior oblique |
| SAE | Severe adverse events |
| SIC | Subject identification code |
| T-bil | Total bilirubin |
| TBV | Total blood volume |
| T-cho | Total cholesterol |
| TG | Triglyceride |
| TOPCARE-AMI | Transplantation of Progenitor Cells and Regeneration Enhancement in<br>Acute Myocardial Infarction |
| T-pro | Total protein |
| VTBI | Volume to be injected |
| WISE | Women's Ischemia Syndrome Evaluation |

| 4, | T | TABLE OF CONTENTS | |
|---|---|---|---|
| 1. | PERSONNEL AND FACILITIES3 | | |
| 2. | STUDY SYNOPSIS4 | | |
| 3. | LIS | T OF ABBREVIATIONS | . 11 |
| 4. | | BLE OF CONTENTS | |
| 5. | SC | HEDULE OF ASSESSMENTS | . 18 |
| 6. | BA | CKGROUND AND SIGNIFICANCE | . 21 |
| | 6.1 | Coronary Microvascular Dysfunction | . 21 |
| | 6.2 | CD34+ Cell Therapy | . 21 |
| | 6.3 | Findings from Nonclinical Studies | |
| | | 6.3.1 Therapeutic Potential of Ex Vivo Expanded Endothelial Progenitor C | ells |
| | | in Myocardial Ischemia in Rats | . 22 |
| | | 6.3.2 Human CD34+ Cell Therapy in Rat Model of Myocardial Ischemia | . 23 |
| | 6.4 | Findings from Clinical Studies | . 23 |
| | | 6.4.1 Intramyocardial Autologous CD34+ Cell Therapy for Refractory Angi | na |
| | | (ACT34-CMI) | . 23 |
| | | 6.4.2 Autologous CD34+ Cell Therapy for Heart Failure | . 24 |
| | 6.5 | Description of Investigational Product | . 25 |
| 7. | ST | UDY OBJECTIVES | . 25 |
| | 7.1 | Primary Objective | . 25 |
| | 7.2 | Secondary Objectives | . 25 |
| 8. | ST | UDY DESIGN | . 26 |
| | 8.1 | Screening Phase | . 26 |
| | 8.2 | Treatment Phase | . 26 |
| | 8.3 | Follow-up Phase | . 27 |
| | 8.4 | Duration of Subject Participation | . 27 |
| | 8.5 | Randomization and Blinding | . 27 |
| | 8.6 | Stopping Rules | . 27 |
| | | 8.6.1 Stopping for Individual Patients | . 27 |
| | | 8.6.2 Stopping of the Study | . 28 |
| 9. | ST | UDY ENDPOINTS | . 28 |
| | 9.1 | Safety Endpoints | . 28 |
| | 9.2 | Efficacy Endpoints | . 28 |
| | 9.3 | Exploratory Cardiac Biomarkers | . 29 |
| 10 | . STI | UDY POPULATION | . 29 |
| | 10.1 | Inclusion Criteria | . 29 |
| | 10 2 | Exclusion Criteria | 30 |

| 11. IN | /ESTIGATIONAL PRODUCT | 31 |
|--------|---------------------------------------------------|----|
| 11.1 | | |
| 11.2 | | |
| 11.3 | Description of Treatment | 32 |
| 11.4 | Investigational Product Accountability | 33 |
| 11.5 | Packaging, Labeling, and Storage | 34 |
| 11.6 | Administration | 34 |
| 11.7 | Completion of CLBS16 product release testing | 35 |
| 11.8 | Procedure for unblinding | 35 |
| 12. ST | UDY VISIT ASSESSMENTS | 35 |
| 12.1 | Screening Visits | |
| 12.2 | Pre-treatment Visits | |
| 12.3 | Treatment Visit (Day 0) | 37 |
| | 12.3.1 Pre-infusion of IP | 37 |
| | 12.3.2 IP infusion (Time 0 hrs) | 37 |
| | 12.3.3 Post-infusion of IP (Time 2, 4, and 6 hrs) | 37 |
| 12.4 | Day 1 visit | 38 |
| 12.5 | Day 8 visit | 38 |
| 12.6 | Day 30 visit | |
| 12.7 | Day 90 Visit | 38 |
| 12.8 | Day 180 visits | 39 |
| | Day 365 visit | 39 |
| 13. SU | BJECT MANAGEMENT | 40 |
| 13.1 | Informed Consent and Enrollment | 40 |
| 13.2 | Subject Identification Code (SIC) | 40 |
| 13.3 | Screening | 40 |
| 13.4 | Randomization | 40 |
| 13.5 | Study Visits | 40 |
| 13.6 | Recording of Medications and Non-Drug Therapies | 41 |
| | Procedures for Monitoring Subject Compliance | |
| 13.8 | Subject Completion/Discontinuation | 41 |
| 14. AS | SESSMENTS OF EFFICACY | 41 |
| 14.1 | ® | 42 |
| 14.2 | | 42 |
| 14.3 | | 42 |
| 14.4 | *************************************** | 42 |
| 14.5 | | 43 |

| 14.6 | Peripheral Arterial Tonometry | 43 |
|--------|---------------------------------------------------|----|
| 14.7 | | 44 |
| 14.8 | Coronary Reactivity Testing | 44 |
| 14.9 | CCS Angina Classification | 45 |
| 15. AS | SESSMENT OF SAFETY | 45 |
| 15.1 | Medical, Medication, and Non-Drug Therapy History | 45 |
| 15.2 | Physical Examinations | 46 |
| 15.3 | Clinical Laboratory Parameters | 46 |
| | 15.3.1 Hematology | 46 |
| | 15.3.2 Clinical Chemistry | 46 |
| | 15.3.3 Lipid Panel | 47 |
| | 15.3.4 Urinalysis | 47 |
| | 15.3.5 Pregnancy Testing | 47 |
| | 15.3.6 Infection Tests | 47 |
| 15.4 | Vital Signs | 47 |
| 15.5 | Adverse Events | 48 |
| | 15.5.1 Serious Adverse Event | 48 |
| | 15.5.2 Non-Serious Adverse Event | 49 |
| | 15.5.3 Adverse Events of Special Interest | 49 |
| | 15.5.4 Severity | 49 |
| | 15.5.5 Causality | 49 |
| | 15.5.6 Reporting for Adverse Events | 50 |
| | 15.5.7 Preexisting Diseases | 51 |
| | 15.5.8 Assessment of Adverse Events | 51 |
| 16. ST | ATISTICS | 52 |
| 16.1 | Sample Size and Power Calculations | 52 |
| 16.2 | Analysis populations | 52 |
| | 16.2.1 Safety analysis set | 52 |
| | 16.2.2 Intent to treat analysis set | |
| | 16.2.3 Per-protocol analysis set | 52 |
| 16.3 | Planned Statistical Analysis | 53 |
| 17. DA | TA HANDLING AND RECORD KEEPING | 53 |
| 17.1 | Confidentiality Policy | 53 |
| | Study Documents | |
| | Document and Data Retention | |
| 17.4 | Direct Access to Source Data/Documents | 54 |

| 18. QU | ALITY CONTROL AND QUALITY A | ASSURANCE | 54 |
|---|---|---|---|
| 18.1 | Investigator's Responsibility | | 54 |
| 18.2 | Investigator Report and Final Clinic | al Study Report | 55 |
| 18.3 | Training | | 55 |
| 18.4 | Auditing | | 55 |
| 18.5 | Non-Compliance with the Protocol . | | 55 |
| 19. ET | HICS | | 56 |
| 19.1 | Compliance Statement | | 56 |
| 19.2 | Participating Centers | | 56 |
| 19.3 | Informed Consent | | 56 |
| 19.4 | Subject Privacy | | 57 |
| 19.5 | Risks and Benefits | | 57 |
| 19.6 | Ethics Committee and Regulatory A | Authorities | 57 |
| 20. ST | UDY ADMINISTRATION | | 58 |
| 20.1 | Monitoring | | 58 |
| 20.2 | Medical Monitor | | 58 |
| 20.3 | Financing and Insurance | | 58 |
| 20.4 | Publication Policy | | 58 |
| 21. SU | PPLEMENTS | | 59 |
| 21.1 | Study Flow Diagram | | 59 |
| 21.2 | Peripheral Arterial Tonometry Work | sheet | 60 |
| 21.3 | | | 64 |
| 21.4 | | | 65 |
| 21.5 | | | 68 |
| 21.6 | | | 72 |
| 21.7 | Invasive Coronary Reactivity Testin | g – Screening and Month 6 | 77 |
| 21.8 | Cell Delivery Protocol | | 82 |
| 22. SIC | SNIFICANT CHANGES FROM PRO | TOCOL VERSION 6 | 83 |
| 23. RE | FERENCES | | 84 |
| INVEST | IGATOR ACKNOWLEDGEMENT | | 89 |

#### 5. SCHEDULE OF ASSESSMENTS





This document and its contents are the property of Caladrius Biosciences, Inc. and are confidential. UNAUTHORIZED COPYING OR USE IS PROHIBITED.



This document and its contents are the property of Caladrius Biosciences, Inc. and are confidential. UNAUTHORIZED COPYING OR USE IS PROHIBITED.





This document and its contents are the property of Caladrius Biosciences, Inc. and are confidential. UNAUTHORIZED COPYING OR USE IS PROHIBITED.

#### 6. BACKGROUND AND SIGNIFICANCE

## 6.1 Coronary Microvascular Dysfunction

Patients with symptoms, evidence of ischemia, and no obstructive coronary artery disease (CAD) are prevalent and increasing in frequency.<sup>3</sup> The prevalence of nonobstructive CAD at coronary angiography amongst patients presenting with chest pain is 20% to 30%<sup>4, 5</sup> and has been reported to be up to 50%.<sup>6</sup> Such patients have disability, healthcare resource consumption, and costs similar to those with obstructive CAD.<sup>7, 8</sup> Functional coronary microvascular abnormalities mediate ischemia and cause angina<sup>9, 10</sup> and have been linked to adverse clinical outcomes.<sup>11, 12</sup> Thus, coronary microvascular dysfunction (CMD) may serve as the underlying mechanism for the symptoms and cardiovascular events observed in patients with nonobstructive ischemic heart disease (IHD).

In a recent study of patients with chest pain and nonobstructive CAD (N=1,439) who underwent a comprehensive and invasive assessment of coronary microvascular function, more than two-thirds of patients had some sort of coronary microvascular dysfunction. 13 Considerable data document that CMD contributes to myocardial perfusion abnormalities in regions supplied by vessels without epicardial stenosis<sup>14, 15, 16</sup> in patients with risk factors and/or angina, but without epicardial stenosis. 17, 18, 19, 20 It is now evident that CMD is not benign and is predictive of adverse cardiovascular outcomes. In the MESA (Multi-Ethnic Study of Atherosclerosis), both myocardial flow (cardiac magnetic resonance imaging [cMRII]) during adenosine-induced hyperemia and flow reserve were inversely associated with risk factor burden.<sup>21</sup> CMD has been documented among symptomatic women without flow-limiting coronary stenosis in the Women's Ischemia Syndrome Evaluation (WISE)<sup>22, 23</sup> by directly measured (Doppler flow wire) coronary flow, by cMRI,<sup>24</sup> and by positron emission tomography (PET),<sup>11</sup> These studies have linked CMD and atherosclerosis risk factors with adverse outcomes over follow-up. CMD has also been replicated in another female cohort.<sup>25</sup> providing additional support for its link with several risk factors.

# 6.2 CD34+ Cell Therapy

The potential role of autologous CD34+ cells for the treatment of CMD is supported by findings from the Doppler Substudy of the REPAIR-AMI trial, which demonstrated that coronary microvascular function improved with administration of progenitor cells in patients with reperfused acute myocardial infarction. Intracoronary infusion of bone marrow cells (BMCs; rich in CD34+ cells) in patients with reperfused AMI was associated with a normalization of CFR in the infarct-related artery within 4 months and hence a profound improvement in maximal vascular conductance capacity. Therefore,

these data support the hypothesis that BMCs infused into the coronary circulation reconstitute damaged endothelium and promote neovascularization in the area of the infarct vessel in patients with acute myocardial infarction (AMI).<sup>26</sup> These results are supported by the Transplantation of Progenitor Cells and Regeneration Enhancement in Acute Myocardial Infarction (TOPCARE-AMI) trial, which was not placebo controlled and suggested that intracoronary transplantation of progenitor cells effectively improves CFR in the infarct-related artery in patients with successfully reperfused AMI.<sup>27</sup>

Intracoronary cell delivery may be applicable to patients with CMD. The efficacy of cell delivery in treatment of cardiovascular disease is gaining interest, and cell therapy with CD34+ cells has been shown to be safe and feasible. While cell therapy has been explored in treatment of late stage coronary atherosclerosis such as acute myocardial infarction, no study to date has evaluated the role of cell therapy in patients with early coronary atherosclerosis, non-obstructive coronary arteries, and CMD.

## 6.3 Findings from Nonclinical Studies

# 6.3.1 Therapeutic Potential of Ex Vivo Expanded Endothelial Progenitor Cells in Myocardial Ischemia in Rats

In a study conducted by Kawamoto *et. al.*, the researchers examined the therapeutic potential and safety of endothelial progenitor cells (EPCs) in an animal model of myocardial ischemia.<sup>28</sup> Peripheral blood MNCs obtained from healthy human adults were cultured to promote the growth of EPCs and injected intravenously (IV) into rat models of myocardial ischemia. Five rats were injected with 1 x 10<sup>6</sup> EPCs 3 hours after ischemia induction (EPC group) and the control group (5 rats) received culture media alone.

Echocardiography, performed at baseline and 28 days after ischemia, revealed ventricular dimensions that were significantly smaller and fractional shortening that was significantly greater in the EPC vs. control group by Day 28. Regional wall motion was better preserved in the EPC vs. control group. Following sacrifice on Day 28, necropsy examination revealed that capillary density was significantly greater in the EPC group than in the control group. Additionally, the extent of left ventricular (LV) scarring was significantly less in rats receiving EPCs compared to the controls. Immunohistochemistry revealed capillaries that were positive for human-specific EPCs.

The conclusion from the study was that *ex vivo* expanded progenitor cells can incorporate into foci of myocardial neovascularization and have a favorable impact on preservation of LV function.

## 6.3.2 Human CD34+ Cell Therapy in Rat Model of Myocardial Ischemia

A safety and efficacy study was performed with human CD34+ cells in the athymic nude rat model of myocardial ischemia.\* Mononuclear cells (MNCs) were collected by apheresis from a healthy human volunteer who underwent mobilization (10 μg/kg G-CSF subcutaneously) 3 days prior to MNC collection. CD34+ cells were isolated and injected into rat models of myocardial ischemia via intramyocardial injection. Animals were assigned to one of 6 treatment groups: phosphate buffered saline (PBS); 5 x 10<sup>3</sup> CD34+ cells/kg; 5 x 10<sup>5</sup> CD34+ cells/kg; 5 x 10<sup>5</sup> unselected MNC; or a high dose unselected MNC group that contained 5 x 10<sup>5</sup> unselected CD34+ cells.

Analysis of the efficacy data revealed a statistically significant improvement in both fractional shortening ( $29.5\pm1.6\%$  vs.  $23.23\pm2.5\%$ , p<0.05) and regional wall motion score ( $22.5\pm0.6$  vs.  $24.4\pm0.7$ , p<0.05) in animals treated with 5 x  $10^5$  CD34+ cells/kg when compared to animals in the PBS group, respectively. A statistically significant improvement was also noted in fractional shortening (FS) ( $28.8\pm1.8\%$  vs.  $23.23\pm2.5\%$ , p<0.05) in animals treated with the high dose of unselected MNC containing 5 x  $10^5$  unselected CD34+ cells when compared to animals treated with PBS.

Moreover, in all animals studied for 28 days, the percent of fibrosis was calculated by morphometric analysis of 4 representative elastic tissue trichrome stained sections for each animal. The percent fibrosis/entire left ventricular area was significantly lower in animals treated with 5 x 10<sup>5</sup> CD34+ cells/kg when compared to animals treated in any other group (15.9±1.5% vs. 23.7±1.4% PBS group, 23.8±2.7 low dose CD34+ group, 27.2±2.4% low dose MNC group, and 22.7±3.1 high dose MNC group, p<0. 03).

The pre-clinical studies above show that EPCs and CD34+ cells are safe and efficacious for myocardial ischemia treatment in the rat model.

## 6.4 Findings from Clinical Studies

# 6.4.1 Intramyocardial Autologous CD34+ Cell Therapy for Refractory Angina (ACT34-CMI)

Losordo et al. conducted a prospective, double-blind, randomized, phase 2 study (NCT00300053) in 167 patients with no-option refractory angina evaluating 2 doses (1x10<sup>5</sup> or 5x10<sup>5</sup> cells/kg) of mobilized autologous CD34+ cells compared with an equal volume of diluent (placebo).<sup>29</sup> Treatment was distributed into 10 sites of ischemic, viable

<sup>\*</sup> Data on file; BB-IND 11196 Pharmacology and Toxicology Section C.

myocardium with a NOGA™ mapping injection catheter. The primary outcome measure was weekly angina frequency 6 months after treatment. Weekly angina frequency was significantly lower in the low-dose group than in placebo-treated patients at both 6 months (6.8±1.1 versus 10.9±1.2, P=0.020) and 12 months (6.3±1.2 versus 11.0±1.2, P=0.035); measurements in the high-dose group were also lower, but not significantly. Similarly, improvement in exercise tolerance was significantly greater in low-dose patients than in placebo-treated patients (6 months: 139±151 versus 69±122 seconds, P=0.014; 12 months: 140±171 versus 58±146 seconds, P=0.017) and greater, but not significantly, in the high-dose group. During cell mobilization and collection, 4.6% of patients had cardiac enzyme elevations consistent with non-ST segment elevation myocardial infarction. Mortality at 12 months was 5.4% in the placebo-treatment group with no deaths among cell-treated patients. These results provide evidence for the potential bioactivity of autologous CD34+ cells in myocardial ischemia as well as demonstrating the feasibility of this treatment strategy in a multi-center study.

## 6.4.2 Autologous CD34+ Cell Therapy for Heart Failure

Vrtovec et al. have performed a prospective, randomized clinical study (NCT01350310) investigating long-term effects of CD34+ stem cell therapy in patients with nonischemic dilated cardiomyopathy (DCM).30 Of 110 patients with DCM, 55 were randomized to CD34+ cell transplantation (SC group) and 55 patients did not receive stem cell therapy (Controls). In the SC group, peripheral blood CD34+ cells were mobilized by granulocyte-colony stimulating factor and collected via apheresis. Patients underwent myocardial scintigraphy, and CD34+ cells were injected in the coronary artery supplying the segments with reduced viability. At 5 years, stem cell therapy was associated with an increase in LVEF (from  $24.3 \pm 6.5\%$  to  $30.0 \pm 5.1\%$ ; P = 0.02), an increase in 6minute walk distance (from 344 ± 90 m to 477 ± 130 m; P < 0.001), and a decrease in Nterminal pro B-type natriuretic peptide (NT-proBNP) (from 2322 ± 1234 pg/mL to 1011 ± 893 pg/mL; P <0.01). During follow-up, 27 (25%) patients died, and 9 (8%) underwent heart transplantation. Of the 27 deaths, 13 were attributed to pump failure and 14 to sudden cardiac death. Total mortality was lower in patients receiving SC therapy (8/55, 14%) than in Controls (19/55, 35%) (P = 0.01). The same was true of the pump failure (3/55 vs. 10/55, P = 0.03) but not of the sudden cardiac death (5/55 vs. 9/55, P = 0.39). Thus, it appears that intracoronary stem cell transplantation is associated with improved ventricular remodeling, better exercise tolerance, and improved long-term survival in patients with chronic heart failure due to nonischemic dilated cardiomyopathy.

In addition, Poglagen, et al. investigated the clinical effects of intramyocardial transplantation of selected CD34+ stem cells in patients with ischemic cardiomyopathy in a prospective Phase 1 crossover study (NCT01350310).<sup>31</sup> A total of 33 patients with

ischemic cardiomyopathy and New York Heart Association class III and left ventricular ejection fraction <40% were enrolled. In phase 1, patients were treated with medical therapy for 6 months. Thereafter, all patients underwent intramyocardial CD34+ cell transplantation. Peripheral blood CD34+ cells were mobilized by granulocyte colony stimulating factor, collected via apheresis, and injected intramyocardially in the areas of hibernating myocardium. Patients were followed up for 6 months after the procedure (phase 2). Two patients died during phase 1 and none during phase 2. The remaining 31 patients were 85% men, aged 57±6 years. In phase 1, we found no change in left ventricular ejection fraction (from 25.2±6.2% to 27.1±6.6%; P=0.23), NT-proBNP (from 3322±3411 to 3672±5165 pg/mL; P=0.75) or 6-minute walk distance (from 373±68 to 411±116 m; P=0.17). In contrast, in phase 2 there was an improvement in left ventricular ejection fraction (from 27.1±6.6% to 34.9±10.9%; P=0.001), increase in 6minute walk distance (from 411±116 to 496±113 m; P=0.001), and a decrease in NTproBNP (from 3672±5165 to 1488±1847 pg/mL; P=0.04). The average number of injected CD34+ cells was 90.6±7.5×106. Higher doses of CD34+ cells and a more diffuse distribution of intramyocardial cell injections were associated with better clinical response. These findings suggest that intramyocardial CD34+ cell transplantation may be associated with improved left ventricular function, decreased NT-proBNP levels, and better exercise capacity in patients with ischemic cardiomyopathy.

## 6.5 Description of Investigational Product

#### STUDY OBJECTIVES

## 7.1 Primary Objective

To evaluate the safety and tolerability of intracoronary delivery of CLBS16 in patients with CMD and without obstructive coronary artery disease.

#### 7.2 Secondary Objectives

To evaluate the potential efficacy of CLBS16 by examining the following exploratory parameters:

Coronary microvascular function as measured by coronary flow reserve



Peripheral arterial tonometry (PAT)



#### STUDY DESIGN

This is a phase 2 open-label clinical study to evaluate the safety, tolerability, and potential bioactivity of CLBS16 in patients with coronary microvascular dysfunction and no obstructive coronary artery disease. The study will be conducted in the phases as outlined below:

## 8.1 Screening Phase

Patients who provide informed consent will be screened for eligibility within 60 days before beginning the study treatment phase. Patients must be on stable medical therapy for 30 days prior to screening and until treatment with CLBS16.



#### 8.2 Treatment Phase





#### 8.3 Follow-up Phase

will be collected for all subjects during the treatment and 12 month follow-up period to evaluate the safety and tolerability of intracoronary administration of CLBS16. Efficacy assessments will be performed through 6 months to evaluate the potential bioactivity of CLBS16 in patients with coronary microvascular dysfunction.



## 8.4 Duration of Subject Participation

All subjects will be followed for 12 months following intracoronary administration of CLBS16.

## 8.5 Randomization and Blinding

This is an open-label study with a single group receiving intracoronary CLBS16 infusion, therefore randomization and blinding do not apply to this clinical study.

# 8.6 Stopping Rules

# 8.6.1 Stopping for Individual Patients

Treatment of an individual patient should not be undertaken if any issue is identified which would create an unreasonable risk for intracoronary administration of CLBS16. Treatment should also not be undertaken if any issue is identified which would create an unreasonable risk for coronary microvascular testing. Any such decision may be made prior to initiation of the treatment procedure or at any point during a microvascular

testing or intracoronary administration procedure. Patients not treated with CLBS16 may be replaced at the discretion of the Sponsor.



## 8.6.2 Stopping of the Study

The investigators and the medical monitor for this study will review adverse events on an ongoing basis and will communicate with each other if any evolving safety signal is perceived. In the event that an evolving safety signal is perceived, the medical monitor may choose to discontinue treatment of further patients. However, observation of patients already treated should continue to the extent possible.

#### STUDY ENDPOINTS

## 9.1 Safety Endpoints

- Adverse events, including serious adverse events
- Laboratory investigations
- Physical examinations
- Vital signs
- Electrocardiographic findings



## 9.2 Efficacy Endpoints

- · Change from baseline in coronary flow reserve at 6 months
- Change from baseline in peripheral arterial tonometry measurements at 6 months





#### 10. STUDY POPULATION



#### 10.1 Inclusion Criteria

Subjects who meet ALL of the following criteria are eligible for this study:

- Men or women age ≥18
- History of effort-induced anginal symptoms and currently experiencing angina at least 3 times per week.

| 3. | No obstructive disease |
|---|---|
| 4. | If subject is of childbearing potential, presents with a negative pregnancy test, and agrees to employ adequate birth control measures for the duration of the study. |
| 5 | Subject is willing and able to comply with the requirements of the protocol |
| | Stable medical therapy for 30 days prior to screening |
| ٠. | etable medical alorapy for or days prior to sersorming |
| 7. | Able to provide signed informed consent |
| 10 | .2 Exclusion Criteria |
| 1. | Myocardial infarction within 90 days |
| 2. | Prior evidence of obstructive heart disease including history of Percutaneous |
| | Coronary Intervention (PCI) and/or Coronary Artery Bypass Grafting (CABG) |
| | Planned percutaneous coronary intervention or CABG |
| 4. | Diagnosis of other specific cardiac disease |
| 7 | Subject currently uses coumadin, |
| | plans to use one of these agents during the time frame of the trial |
| | Toward by the cold of colde against dening the mile manner of the cold |

11. Subject tests positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C
12. Subject has active inflammatory disease or autoimmune disease, or is in a chronic immunosuppressive state
13. Recent history of abuse or current abuser of recreational drugs
14. Subject is pregnant or lactating
15. Malignant neoplasm

within 5 years prior to screening
16. Subject has participated in another clinical study within 90 days
17. History of sickle cell disease

#### 11. INVESTIGATIONAL PRODUCT

The process for obtaining autologous CD34+ cells is as follows:



The dose level was selected based on results from previous clinical studies, which were able to demonstrate efficacy from intracoronary administration of CD34+ cells. Three studies provide support for the dose level in this study. The first is a study by Leziac, et al. in which it was demonstrated that treatment with CD34+ cells led to improved myocardial perfusion in patients with nonischemic dilated cardiomyopathy.<sup>34</sup> In that study, the maximum dose that could be manufactured was administered, with a range between 54 x 106 cells and 284 x 106 cells. All doses were well tolerated. In a second study, Wang, et al. examined CD34+ cell therapy in patients with intractable angina.35 In their study, the mean number of CD34+ cells infused was also limited by the number of cells available from the manufacturing procedure and averaged 56 ± 23 x 106 cells per patient. In the Wang study, significant improvements were observed in frequency of angina episodes, nitroglycerin use, and other measures. All treatments were well tolerated. The third reference study for cell dose was the study by Vrtovec, et al., in which effects of CD34+ cells were examined in patients with nonischemic dilated cardiomyopathy.30 In that study, the number of cells infused was also limited by the number of cells available from the manufacturing procedure and averaged 113 ± 26 x 10<sup>6</sup> cells per patient. Significant improvements were seen in left ventricular ejection fraction, 6 minute walk test, and other measures out to 5 years after treatment. All treatments were well tolerated.

Regarding route of administration, many previous studies have used either intramyocardial injection or intracoronary infusion of CD34+ cells. Both routes of administration have been effective at improving cardiac function. However, there has been no clear evidence that one would be more effective than the other, and due to the less invasive nature of intracoronary infusion versus intramyocardial injection, the intracoronary infusion route of administration was selected.



# 11.4 Investigational Product Accountability

The investigator will ensure that the investigational product (IP) is stored as instructed in the investigational product manual and that the storage area is secured, with access limited to authorized study personnel. The investigator will maintain records that the IP was received, including the date received, IP lot number, date of manufacture or expiration date, amount received, and disposition. IP must be dispensed only at the institution specified for each study site. Records will be maintained that include the subject's initials and subject identification code (SIC), dispensation date, and amount dispensed. All remaining partially used and/or unused IP will be destroyed in accordance with applicable laws and study site procedures or, if requested, returned to the Sponsor or Sponsor's representative. If IP is to be destroyed, the investigator will provide documentation in accordance with Sponsor's specifications.

## 11.5 Packaging, Labeling, and Storage

A label will include subject identifiers, product expiration date & time, clinical site designator, product volume, product identifier, temperature requirements, contact information, processing site information, and applicable cautions and warnings. The cell product is sealed in a doubly wrapped sterile bag and placed in a secure transportation box to be delivered to the cardiac catheterization facility,

#### 11.6 Administration

Upon notification from the cell processing facility that the CLBS16 cell product has been released for infusion (by email), the subject will undergo cardiac catheterization.

The subject will receive standard post cardiac procedure care including repeated examinations of vascular access site for hematomas or local access related complications or retroperitoneal bleed. Subjects will be monitored for 24 hours for

complications, including arrhythmia, ischemia and bleeding from the catheter insertion site.



## 11.8 Procedure for unblinding

This is an open label study so a procedure for unblinding is not applicable.

#### 12. STUDY VISIT ASSESSMENTS



At the first screening visit, perform the following:

- Administer informed consent
- Perform peripheral arterial tonometry
- Review inclusion and exclusion criteria to determine study eligibility
- Collect medical history including demographics (i.e. gender, date of birth, race, and ethnicity)
- Collect information on concomitant medications (including non-drug therapies)
- · Assess for adverse events
- Perform physical examination
- •
- Collect vital signs
- Collect blood for hematology and clinical chemistry

- Collect blood for lipid panel
- Collect urine and perform urinalysis
- Collect blood and perform infection tests (including HIV antibody, HBs antigen, HBc antibody, and HCV antibody)
- Perform urine pregnancy test on female subjects of childbearing potential
- Perform 12-lead ECG



At the second screening visit, perform the following:

- Perform coronary angiography and coronary microvascular testing if needed (see Supplement 21.7; may be performed on a different day if needed)
- Assess for adverse events
- Collect information on concomitant medications (including non-drug therapies)
- Review inclusion and exclusion criteria to confirm study eligibility

# 12.2 Pre-treatment Visits

The following will be performed or assessed at each of the pre-treatment study days unless noted:

- Collect information on concomitant medications (including non-drug therapies)
- Assess for adverse events
- Review inclusion and exclusion criteria to confirm study eligibility
- Perform vital signs
- Perform urine pregnancy test on female subjects of childbearing potential (only on pre-treatment Day 1)
- Perform 12-lead ECG (only on pre-treatment Day 1)
- Collect blood for hematology



### 12.3 Treatment Visit (Day 0)

#### 12.3.1 Pre-infusion of IP

The following will be performed or assessed approximately 2 hours prior to infusion:

- Collect information on concomitant medications (including non-drug therapies)
- Assess for adverse events
- Perform targeted physical exam
- Collect blood for hematology and clinical chemistry
- Perform urine pregnancy test on female subjects of childbearing potential
- Perform vital signs
- Perform 12-lead ECG
- · Confirm eligibility criteria prior to IP infusion
- If applicable, admit for overnight hospitalization (subjects may be monitored overnight in the hospital at the discretion of the investigator)

# 12.3.2 IP infusion (Time 0 hrs)

- · Perform vital signs prior to infusion
- Perform intracoronary infusion of IP
- Assess for adverse events

# 12.3.3 Post-infusion of IP (Time 2, 4, and 6 hrs)

The following will be performed or assessed approximately 2, 4, and 6 hours post IP infusion:

- Perform vital signs
- · Perform 12-lead ECG (only at the 2 and 6 hour time points)
- Assess for adverse events

### 12.4 Day 1 visit

- Collect information on concomitant medications (including non-drug therapies)
- Perform vital signs
- Perform 12-lead ECG
- Collect blood for hematology and clinical chemistry
- Assess for adverse events
- Discharge from hospital, if applicable

## 12.5 Day 8 visit

adverse events and concomitant medications including non-drug therapies.

- Collect information on concomitant medications (including non-drug therapies)
- Assess for adverse events

## 12.6 Day 30 visit

- Collect information on concomitant medications (including non-drug therapies)
- · Perform vital signs (only if patient makes in person visit)
- Collect blood for hematology and clinical chemistry

- Assess for adverse events
- , leaded for dateled events

# 12.7 Day 90 Visit

collect information on adverse events and concomitant medications including non-drug therapies. Additionally, the site will have provided

- Collect information on concomitant medications (including non-drug therapies)
- Perform vital signs (only if patient makes in person visit)
- Assess for adverse events

### 12.8 Day 180 visits

Also note that these procedures may be performed across more than one visit day, within a span of 7 days.



Perform peripheral arterial tonometry



- Collect information on concomitant medications (including non-drug therapies)
- Assess for adverse events
- Perform 12-lead ECG
- Perform vital signs
- Collect blood for hematology and clinical chemistry
- Collect blood for lipid panel
- Perform targeted physical exam
- Perform coronary angiography and coronary microvascular testing
- Perform pregnancy test on females of childbearing potential

# 12.9 Day 365 visit

The subject will receive a phone call from the investigative site to collect information on adverse events and concomitant medications including non-drug therapies.

### 13. SUBJECT MANAGEMENT

#### 13.1 Informed Consent and Enrollment

Subjects will be enrolled when they have provided informed consent (i.e., signs and dates the informed consent form to participate in the study), met all inclusion and none of the exclusion criteria, and completed the screening phase.

### 13.2 Subject Identification Code (SIC)

The following series of numbers will comprise the SIC: protocol number (e.g., CLBS16-P01), 3-digit number study site number (e.g., 002) to be provided by the Sponsor, and 3-digit subject number (e.g., 003) reflecting the order of enrollment (i.e., signing the informed consent form). For example, the third subject who signed an informed consent form at study site 002 will be identified as Subject CLBS16-P01-002-003. All study documents [e.g., clinical documentation, sample containers, drug accountability logs, etc.] will be identified with the SIC.

### 13.3 Screening

Subjects must provide informed consent and meet all inclusion/exclusion criteria and have screening procedures performed within the screening window
Subjects who have failed the screening process will be recorded as a screen failure.
The study site is responsible for maintaining a screening/enrollment log that includes all subjects evaluated for inclusion in the study. The log also will serve to document the reason for screening failure. All screening data will be collected and reported, regardless of screening outcome.

Re-screening of subjects is allowed, at the discretion of the investigator with prior approval from the study Sponsor, unless there are clinical implications that impact the ability of subject to meet selection criteria change.

#### 13.4 Randomization

This is an open-label study with a single group receiving intracoronary CLBS16 infusion, therefore randomization and blinding do not apply to this clinical study.

### 13.5 Study Visits

The overall study design is illustrated in Supplement 21.1, Study Flow Diagram. Details on the procedures to be performed at each study visit, including screening, can be found in Section 5. Detail of procedures performed at each study visit can be found in Section 12.

### 13.6 Recording of Medications and Non-Drug Therapies

Beginning from the time of consent, all medications taken and non-drug therapies received and all concomitant medications taken or administered during the study will be documented in the subject's study records.

### 13.7 Procedures for Monitoring Subject Compliance

All study procedures are to be performed by the investigator or under his/her designation to a co-investigator or study team member, and thus, no separate procedures will be used to monitor subject compliance.

### 13.8 Subject Completion/Discontinuation

A subject is considered to have completed the study when he/she ceases active participation in the study because the subject has, or is presumed to have, followed the protocol. Reasons for completion/discontinuation will be reported, including: completed, screen failure, adverse event (e.g., death), discontinuation by subject (e.g., lost to follow-up [defined as 3 documented unsuccessful attempts to contact the subject], dropout), physician decision (e.g., pregnancy, progressive disease, non-compliance with IP/protocol violation(s), recovery), study terminated by Sponsor, or other (reason to be specified by the investigator, e.g., technical problems). As the IP is administered once on the treatment day, subject will be considered as discontinued from the study only if the subject is unable to cooperate with study visits and study measurements. All data available for the subject up to the time of completion/discontinuation should be recorded.

The reason for discontinuation will be recorded, and data collected up to the time of discontinuation will be used in the analysis and included in the clinical study report.

Subjects withdrawn or discontinued prior to assessment of efficacy at month 6 may be replaced at the discretion of the Sponsor.

For any subject discontinuation or withdrawal, an attempt will be made to obtain followup data, per protocol, through the intended completion of the study, if possible.

#### 14. ASSESSMENTS OF EFFICACY

Note that the efficacy assessments should generally be conducted in the order listed here,





### 14.6 Peripheral Arterial Tonometry

Peripheral arterial tonometry (PAT) will be measured according to the method used by Suessenbacher, et al. 44 PAT should be measured in the fasting state (at least 12 hours). Vasoactive drugs should be withheld since bed time on the previous day. Patients are to be asked not to smoke on the day of the examination. Peripheral endothelial function will be assessed using the commercially available EndoPAT device (Itamar Medical Ltd. Caesarea, Israel). With this device, a beat-to-beat plethysmographic record of the finger arterial pulse wave amplitude is captured using pneumatic probes placed on the index finger of each hand. For the assessment of endothelial function, the reactive hyperemia technique is to be used. Measurements are to be obtained for 6 minutes at baseline (at rest) followed by 5 minutes of occlusion of the right upper arm with a sphygmomanometer cuff inflated to a suprasystolic level (50 mm Hg above the initially measured systolic blood pressure). The cuff is then deflated to induce reactive (flowmediated) hyperemia, which is measured for 5 or more minutes. The left hand remains unoccluded as a reference to correct for systemic changes. The PAT-ratio, which represents endothelial function, is calculated as the ratio between the magnitude of the average postocclusive pulse wave amplitude (1.5 to 2.5 minutes after the release of arterial occlusion) and the average pulse wave amplitude observed over 6 minutes of preocclusion, corrected for systemic changes. A worksheet for PAT measures is provided in Supplement 21.2.



### 14.8 Coronary Reactivity Testing

A detailed description of the coronary reactivity testing is found in Supplement 21.7.



#### 15. ASSESSMENT OF SAFETY

# 15.1 Medical, Medication, and Non-Drug Therapy History

At screening, the subject's medical history will be described for the following body systems including past surgeries and start and end dates, if known: eyes, ears, nose, and throat; respiratory; cardiovascular; gastrointestinal; musculoskeletal; neurological; endocrine; hematopoietic/lymphatic; dermatological; and genitourinary.

All medications taken and non-drug therapies received from the signing of informed consent until completion/termination will be recorded as concomitant medications and non-drug therapies.

Concomitant medications in general are allowed broadly except in cases where they might represent a hazard for the patient or be indicative of an underlying condition that would put the patient at risk.

# 15.2 Physical Examinations

At screening and subsequent study visits, a physical examination will be performed. A complete physical exam assessment includes general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological. Targeted physical examinations will be symptom-directed. The physical examinations should be performed by the same investigator each time, whenever possible. If an abnormal condition is detected at screening, the condition will be described on the medical history form. At subsequent study visits, if a new abnormal or worsened abnormal pre-existing condition is detected, the condition will be described on the AE form.

### 15.3 Clinical Laboratory Parameters

### 15.3.1 Hematology

The hematology panel will consist of complete blood count (hemoglobin, hematocrit, erythrocytes [i.e., red blood cell count], and leukocytes [i.e., white blood cell count]) with differential (i.e., basophils, eosinophils, lymphocytes, monocytes, neutrophils), platelet counts, prothrombin time (PT; sec) or international normalized ratio (INR), and activated partial thromboplastin time (APTT; sec). A limited hematology assessment will be performed on pre-treatment visit days and at the Treatment Visit (Day 0), which will only include the complete blood count (CBC) with differential, and platelet counts. Hematology can be evaluated in either the fed or fasted state.

### 15.3.2 Clinical Chemistry

The clinical chemistry panel will consist of creatinine, estimated glomerular filtration rate (e-GRF), creatine kinase (CK), electrolytes (sodium, potassium, chloride, calcium, magnesium, and phosphate), bicarbonate, total protein (T-pro), albumin, alanine aminotransferase (ALT), total bilirubin (T-bil), alkaline phosphatase (ALP), aspartate aminotransferase (AST), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and glucose. If hsCRP is not collected as part of cardiac biomarkers, the C-reactive protein

(CRP) should be collected as part of clinical chemistry. Clinical chemistry will be evaluated in the fasted state.

### 15.3.3 Lipid Panel

The lipid panel will consist of total cholesterol (T-cho), high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglyceride (TG). It will be evaluated in the fasted state.

### 15.3.4 Urinalysis

The urinalysis panel will consist of protein, occult blood, glucose, urobilinogen, bilirubin, ketones, and sediments.

### 15.3.5 Pregnancy Testing

Urine pregnancy testing for human chorionic gonadotrophin (hCG) will be performed on females of childbearing potential.

### 15.3.6 Infection Tests

The following infection tests will be performed: HBs antigen, HBc antibody, HCV antibody, and HIV antibody.

### 15.4 Vital Signs

Vital signs will include body temperature (°F), respiratory rate (breaths/min), pulse rate (beats/min), systolic and diastolic blood pressure (mm Hg), height (in or cm, only at the screening visit) and weight (lb or kg). Blood pressures should be measured in the sitting position after 5 minutes of rest. Vital signs will be measured at screening, during the Pre-Treatment Period, within 30 minutes before and after administration of IP on Day 0, and at each study visit and at study completion/termination. Vital signs will be collected at Day 90 only if the patient makes an in-person visit. Additionally, blood pressure and pulse rate will be monitored at the following timepoints (these will not be made part of the clinical database):

- Within 30 minutes before apheresis and approximately every 15 minutes during apheresis
- Pulse rate and blood pressure will be monitored approximately every 15 minutes during cardiac catheterization

Vital sign values are to be recorded. For each vital sign value, the investigator will determine whether the value is considered an AE (see definition in Section 15.1). If

assessed as an AE, the medical diagnosis (preferably), symptom, or sign will be recorded on the AE form. Additional tests and other evaluations required to establish the significance or etiology of an abnormal result or to monitor the course of an AE should be obtained when clinically indicated. Any abnormal value that persists should be followed at the discretion of the investigator.

#### 15.5 Adverse Events

All AEs will be recorded from signing the informed consent until study completion or discontinuation. An AE is defined as any untoward medical occurrence in a subject administered IP, regardless of a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of an IP, whether or not related to the IP. An AE includes any event, regardless of the presumed causality between the event and the IP.

Any subject experiencing an AE will be examined by a physician as soon as possible. The physician in attendance will do whatever is medically necessary for the safety and well-being of the subject. The subject will remain under observation as long as medically indicated in the opinion of the investigator. Non-serious AEs will be followed until the end of subject participation in the study.

#### 15.5.1 Serious Adverse Event

A adverse event is considered serious if, in the view of either the investigator or the Sponsor, it results in any of the following outcomes:

- Outcome is fatal/results in death
- Is life-threatening (at the time of the event)
- Requires hospitalization or results in prolongation of an existing hospitalization
- Results in persistent or significant disability/incapacity
- Results in congenital anomaly/birth defect
- Is a medically important event that may not be immediately life-threatening or require hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the definitions above (e.g., infection, allergic reaction, etc.)

Each Serious Adverse Event (SAE) will be followed until resolution, medically stabilized, or 30 days after end of study visit, whichever comes first. All SAEs are to be reported to the Sponsor within 24 hours of becoming aware of the event.

#### 15.5.2 Non-Serious Adverse Event

A non-serious AE is an AE that does not meet the criteria of a SAE.

### 15.5.3 Adverse Events of Special Interest

The following two adverse events of special interest (AESI) will be collected and tracked in this study:

- Infusions prematurely stopped or paused due to an adverse event
- Infusion-related reactions resulting in discontinuation of infusion or requiring medical treatment

### 15.5.4 Severity

The investigator will assess the severity of each AE using his/her clinical expertise and judgment based on the most appropriate description below:

#### Mild

- The AE is a transient discomfort and does not interfere in a significant manner with the subject's normal functioning level.
- The AE resolves spontaneously or may require minimal therapeutic intervention.

#### Moderate

- The AE produces limited impairment of function and may require therapeutic intervention.
- The AE produces no sequelae.

#### Severe

- The AE results in a marked impairment of function and may lead to temporary inability to resume usual life pattern.
- The AE produces sequelae, which require (prolonged) therapeutic intervention.

### 15.5.5 Causality

Causality is a determination of whether there is a reasonable possibility that the IP is etiologically related to/associated with the AE. Causality to both the IP as well as to the infusion procedure will be assessed. Causality assessment includes, e.g., assessment of temporal relationships, dechallenge/rechallenge information, association (or lack of association) with underlying disease, presence (or absence) of a more likely cause, and physiological plausibility. For each AE, the investigator will assess the causal

relationship between the IP and the AE using his/her clinical expertise and judgement according to the following most appropriate algorithm for the circumstances of the AE:\*

- Not related (both circumstances must be met)
  - Is due to underlying or concurrent illness, complications, concurrent treatments, or effects of concurrent drugs
  - Is not related to the IP (i.e., does not follow a reasonable temporal relationship to the administration of IP or has a much more likely alternative etiology).
  - No rational exists for relatedness
- Unlikely related (either 1 or both circumstances are met)
  - Has little or no temporal relationship to the IP
  - A more likely alternative etiology exists
  - Some (perhaps weak) rational exits for a relatedness
- Possibly related (both circumstances must be met)
  - Follows a reasonable temporal relationship to the administration of IP
  - An alternative etiology is equally or less likely compared to the potential relationship to the IP
- Probably related (both circumstances must be met)
  - Follows a strong temporal relationship to the administration of IP
  - Another etiology is unlikely or significantly less likely
- Definitely related
  - The evidence provides convincing proof of a relationship to the IP

# 15.5.6 Reporting for Adverse Events

All AEs will be recorded from signing the informed consent until study completion or discontinuation. AEs that occur prior to treatment will be considered non-treatment emergent AEs. AEs that occur during or after treatment will be considered treatment emergent AEs. Treatment emergent AEs will be analyzed separately. All AEs will be described using the sign, symptom, or medical diagnosis on the AE form in standard medical terminology in order to avoid the use of vague, ambiguous, or colloquial expressions. Each AE will be defined as a SAE or non-serious AE according to the definitions in Section 15.5.1 and Section 15.5.2, respectively. The investigator will evaluate the severity of each AE and the causal relationship of the event to the administration of study product (see Section 15.5.4 and Section 15.5.5, respectively). The outcome and action taken also will be recorded on the AE form. Non-serious AEs

<sup>\*</sup> From CTC-AE version 4.03

will be followed until the end of subject participation in the study. SAEs will be followed until medically stabilized or 30 days after termination visit, whichever occurs first.



The investigator shall comply with local Food and Drug Administration (FDA) regulations Code of Federal Regulations Title 21 Section 312 [21CFR 312] and any applicable guidance for reporting any SAEs.

### 15.5.7 Preexisting Diseases

Preexisting diseases that are present before entry into the study (as described in the medical history) will not be recorded as AEs but will be documented in the subject initial history. Preexisting diseases that manifest with the same severity, frequency, or duration after IP exposure also will not be recorded as AEs but will be documented in the subject initial history. However, when there is an increase in the severity or duration of a preexisting disease, the event must be described as an AE, and recorded on the form.

#### 15.5.8 Assessment of Adverse Events

Each AE will be described on the AE form using the medical diagnosis (preferred), symptom, or sign, in standard medical terminology in order to avoid the use of vague, ambiguous, or colloquial expressions. Each AE will be evaluated by the investigator for:

- Seriousness as defined in Section 15.5.1 and Section 15.5.2
- Severity as defined in Section 15.5.4
- Causal relationship to IP exposure or study-related procedure as defined in Section 15.5.5

For each AE, the outcome (i.e., recovering/resolving, recovered/resolved, recovered/resolved with sequelae, not recovered/not resolved, fatal) and action taken

will also be recorded on the AE form. Recovering/resolving AEs will be followed until resolution, medically stabilized, or 30 days after the patient's termination visit, whichever comes first.

#### 16. STATISTICS

### 16.1 Sample Size and Power Calculations

This is an exploratory study to estimate the effect of CLBS16 treatment in this population of patients. The primary endpoint of the change in CFR from baseline (screening measurement) to 6 months after treatment will be measured to estimate the



### 16.2 Analysis populations

### 16.2.1 Safety analysis set

The safety analysis set will consist of all subjects who have been consented in the study



### 16.2.2 Intent to treat analysis set

The intent-to-treat analysis (ITT) set will consist of all subjects who received treatment with CLBS16.

## 16.2.3 Per-protocol analysis set

The per-protocol analysis set will exclude subjects who had deviations that may impact critical efficacy variables.

### 16.3 Planned Statistical Analysis

The primary measurements of CFR will be used to estimate the efficacy of treatment and the overall analysis framework will be paired t tests using baseline and 6-month visit data.



### 17. DATA HANDLING AND RECORD KEEPING

### 17.1 Confidentiality Policy

The investigator will comply with the confidentiality policy as described in the Clinical Study Agreement and with national, local, and institution-specific patient privacy regulations.

# 17.2 Study Documents

The investigator will maintain complete and accurate study documentation in a separate file. Documentation may include medical records, records detailing the progress of the study for each subject, signed informed consent forms, drug disposition records, correspondence with the IRB and the study monitor/Sponsor, enrollment and screening information, data worksheets, SAE laboratory reports (if applicable), data clarifications requested by the Sponsor, etc.

The investigator will comply with the procedures for data recording and reporting. Any corrections to study documentation must be performed as follows: 1) the first entry will be crossed out entirely, remaining legible; and 2) each correction must be dated and initialed by the person correcting the entry and include the reason for change, if not obvious. The use of correction fluid and erasing are prohibited.

Questions or interpretations of the protocol will be referred to the Sponsor. The Sponsor is responsible for providing interpretation of all data questions.

Page 54 of 89 26 August 2019

It is recommended that data worksheets be completed within 48 hours of data becoming available

The investigator is responsible for the procurement of data and for the quality of data. Only designated study site personnel shall record or change data. Each correction will require documentation of the reason for the change.

Any data correction will be noted, including old and new values, initials, and date when authorized study personnel made the change.

#### 17.3 Document and Data Retention

The investigator will retain study documentation and data (paper and electronic) in accordance with 21 CFR §312.57 (for 2 years after a marketing application is approved for the drug or until 2 years after the CLBS16 IND has been deactivated, whichever occurs first) and other applicable national, local, and regional regulatory requirements.

#### 17.4 Direct Access to Source Data/Documents

The investigator/study site will cooperate and provide direct access to study documents and data, including source documentation for monitoring by the study monitor, audits by the Sponsor or Sponsor's representatives, review by the IRB, and inspections by applicable regulatory authorities, as described in the Clinical Study Agreement. If contacted by an applicable regulatory authority, the investigator will notify the Sponsor of contact, cooperate with the authority, provide the Sponsor with copies of all documents received from the authority, and allow the Sponsor to comment on any responses, as described in the Clinical Study Agreement.

#### 18. QUALITY CONTROL AND QUALITY ASSURANCE

### 18.1 Investigator's Responsibility

The investigator will comply with the protocol (which has been approved/given favorable opinion by an Institutional Review Board [IRB]), International Council on Harmonisation (ICH), Good Clinical Practice (GCP), and applicable regulatory requirements as described in the Clinical Study Agreement. The investigator is ultimately responsible for the conduct of all aspects of the study at the study site and verifies by signature the integrity of all data transmitted to the Sponsor. The term "investigator" as used in this

protocol and in study documents refers to the investigator or authorized study personnel that the investigator has designated to perform certain duties. Sub-investigators or other authorized study personnel are eligible to sign for the investigator, except where the investigator's signature is specifically required.

### 18.2 Investigator Report and Final Clinical Study Report

The investigator will submit a written report of the study's status to the Sponsor, as described in the Clinical Study Agreement. The investigator will also submit interim progress reports to the Sponsor on a regular basis, as requested.

### 18.3 Training

The study monitor will ensure that the investigator and study site personnel understand all requirements of the protocol, the investigational status of the IP, and his/her regulatory responsibilities as an investigator. Training may be provided at an investigator's meeting, at the study site, and/or by instruction manuals. In addition, the study monitor will be available for consultation with the investigator and will serve as the liaison between the study site and the Sponsor.

### 18.4 Auditing

The Sponsor and/or Sponsor's representatives may conduct audits to evaluate study conduct and compliance with the protocol, standard operating procedures, other written instructions/agreements, ICH GCP, and applicable regulatory guidelines/requirements. The investigator will permit auditors to visit the study site, as described in the Clinical Study Agreement. Auditing processes specific to the study will be described in the auditing plan.

# 18.5 Non-Compliance with the Protocol

The investigator may deviate from the protocol to eliminate an apparent immediate hazard to the subject or when the change(s) involves only logistical or administrative aspects of the study (e.g., change of study monitor, change of phone number). In the event(s) of an apparent immediate hazard to the subject, the investigator will notify the Sponsor immediately by phone and confirm notification to the Sponsor in writing as soon as possible, but within 5 working days after the change is implemented. The investigator will also notify the IRB of the emergency change.

If monitoring and/or auditing identify serious and/or persistent non-compliance with the protocol, the Sponsor may terminate the investigator's participation. The Sponsor will notify the IRB and applicable regulatory authorities of any investigator termination.

#### 19. ETHICS

### 19.1 Compliance Statement

This study will be conducted in accordance with this protocol, the International Council on Harmonisation Guideline for Good Clinical Practice E6(R2) (09 November 2016), Title 21 of the US Code of Federal Regulations (US CFR), and other applicable national and local regulatory requirements.

### 19.2 Participating Centers

Participating clinical sites must have an appropriate IRB governance since they are actively engaged in research and provide informed consent. Health Insurance Portability and Accountability Act (HIPAA) and applicable local regulations will be followed by each participating institution in accordance with each institution's requirements. The participating sites will obtain approval from their corresponding review boards in accordance with their local procedures and institutional requirements.

The investigator is required to keep accurate records to ensure the conduct of the study is fully documented.

The investigational sites participating in this study will maintain the highest degree of confidentiality permitted for the clinical and research information obtained from participants participating in this study. Unless required by the laws permitting copying of records, only the coded identity associated with documents or other participant data may be copied (obscuring any personally identifying information). Authorized representatives, as noted above, are bound to maintain the strict confidentiality of medical and research information that may be linked to identify individuals. The investigational site will normally be notified in advance of auditing visits.

#### 19.3 Informed Consent

Written informed consent will embody the elements of informed consent as described in the Declaration of Helsinki and the ICH Guidelines for GCP and will be in accordance with all applicable laws and regulations. Investigators will enroll patients according to the study eligibility criteria and in compliance with 21 CFR §50 and/or 45 CFR §46. The investigator will exercise no selectivity so that no bias is introduced from this source.

All patients must sign an informed consent form before entering into the study according to applicable regulatory requirements and ICH GCP. Before use, the informed consent form will be reviewed by the Sponsor and approved by an IRB. The informed consent form will include a comprehensive explanation of the proposed treatment without any exculpatory statements, in accordance with the elements required by 21 CFR §50 and/or 45 CFR §46, ICH GCP, and applicable regulatory requirements. Patients will be allowed sufficient time to consider participation in the study. By signing the informed consent form, patients agree that they will complete all evaluations required by the study, unless they withdraw voluntarily or are terminated from the study for any reason.

The Sponsor will provide to the investigator in written form any new information that significantly bears on the subjects' risks associated with IP exposure and study procedures. The informed consent will be updated, if necessary. This new information and/or revised informed consent form, that has been approved by the applicable IRB, will be provided by the investigator to the subjects who consented to participate in the study and are still actively participating.

### 19.4 Subject Privacy

The investigator will comply with applicable subject privacy regulations/guidance as described in the Clinical Study Agreement.

#### 19.5 Risks and Benefits

The risks of this study are presented in the Investigator's Brochure and the informed consent form. There is no guaranteed benefit to subjects for their participation in the study.

# 19.6 Ethics Committee and Regulatory Authorities

Before enrollment of patients into this study, the protocol, informed consent form, any promotional material/advertisements, and any other written information to be provided to the patients will be reviewed and approved/given favorable opinion by an IRB. The Investigator's Brochure will be provided for review. The IRB's composition or a statement that the IRB's composition meets applicable regulatory criteria will be documented. The study will commence only upon the Sponsor's receipt of approval/favorable opinion from the IRB, as described in the Clinical Study Agreement.

If the protocol or any other information given to the subject is amended, the revised documents will be reviewed and approved/given favorable opinion by the IRB. The protocol amendment will only be implemented upon the Sponsor's receipt of approval

and, if required, upon the Sponsor's notification of applicable regulatory authority(ies) approval.

#### 20. STUDY ADMINISTRATION

### 20.1 Monitoring

Throughout the course of the study, the study monitor will make frequent contacts with the investigator. This will include telephone calls and on-site visits. The study will be routinely monitored to ensure compliance with the study protocol and the overall quality of data collected. During the on-site visits, the collected data will be reviewed for completeness and adherence to the protocol. As part of the data audit, source documents will be made available for review by the study monitor. The study monitor may periodically request review of the investigator study file to assure the completeness of documentation in all respects of clinical study conduct.

The study monitor will verify that each patient has proper consent documentation from the patient and/or patient's authorized representative for study procedures and for the release of medical records. The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of regulatory agencies.

On completion of the study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

#### 20.2 Medical Monitor

All adverse events will be recorded on the adverse event forms, and the treatment related SAEs will be sent to the IRB, per their reporting requirements, and to the Sponsor. The study medical monitor or designee will review all adverse event reports. Further details are captured in the study medical monitoring plan.

### 20.3 Financing and Insurance

The investigator will comply with investigator financing, investigator/Sponsor insurance, and subject compensation policies, if applicable, as described in the Clinical Study Agreement.

# 20.4 Publication Policy

The investigator will comply with the publication policy as described in the Clinical Study Agreement.

### 21. SUPPLEMENTS

### 21.1 Study Flow Diagram



# 21.2 Peripheral Arterial Tonometry Worksheet

| Patient ID: | Patient Initials |
|---|---|
| Date:// Time: | : Dominant Arm: Right 🗆 Left 🗆 |
| Sex: Male ☐ Female ☐ Age: _ | Arm Occluded (non-dominant): Right □ Left |
| Room Temp:°F @ begin | ning of test |
| Blood pressure #1/ | _(mm Hg) HR (beats/min) |
| Blood pressure #2 (if necessary) _ | / (mm Hg) HR (beats/min) |
| screen turned away from particle Accessories: micropore tape Environment check: o Temperature 70-75°F | e, thermometer, armrest, blood pressure cuff F, pt 20 minute acclimatization, no breeze obile phones off, patient should avoid talking during |
| cold/warm water), remove je clothing, finger nails trimme Explain test to patient: 20 m uncomfortable, after occlusi Place subject in supine pos Measure patient blood present too tight Ask subject to refrain from ranything Insert patient details: ID, ag | |

#### Assemble:

- □ Probes assembly: (connect a new set of probes to the tubes)
  - Click "Deflate"
  - 2. Insert probe into groove in the arm-support
  - Select finger (preferably the index finger. Very large fingers use little finger; use same finger on both hands)
  - Apply probes: insert test finger into DEFLATED probe (make sure to align the top of the finger with the probe and connector; finger-tip must reach all



the way to the end of the probe).

- 5 Click "Inflate"
- After inflation is completes the finger with the probe attached can be removed from the groove.
- Apply blue foam anchors on the adjacent finger (tubes should not cross) and push to the root of the finger.
- Secure tube by taping the free end in an "S" shape to maintain anchor perpendicular to finger axis.

### □ Reposition patient:

- The forearm should be placed on the Arm-support palm-side down
- The hand should be placed over the edge of the support so the fingers dangle freely.

The probe should not touch:

- Adjacent finger
- Foam anchor
- Thumb
- Arm support
- Anything



### Testing:

□ Pre-recording/Signal Quality

- 1. Click "Standby"
- 2. Adjust gain for optimal signal view
- 3. Inspect signal quality for 1-2 minutes
- Tap on designated occluded (arm with BP cuff) to determine Probe 1 and Probe 2
- Make sure there are no leaks for at least 1 minute, refrain from talking to patient and other staff



#### Please take note of:

mm Hg and not above 300.

Start countdown clock icon in the menu bar

Check the signal of the test arm for incomplete occlusion

| | Screen: After good signal strength for at least 1 minute |
|---|---|
| | Nothing should touch the probe during the test |
| | A recording signal icon should appear pointing at the hard drive |
| Phase | e 1—Baseline |
| | Click "Go" |
| | o Baseline start time: : : |
| | Record for 6 minutes before occlusion |
| | If leaks or problems occur during the baseline; it is still OK to stop the study, replace probes and start over. |
| | Just before occlusion |
| | Adjust gain of designated occluded arm to 20,000 |
| | Inform patient that you are about to occlude for 5 minutes. |
| Phase | 2 - Occlusion |
| | Occlusion Recording 5 minutes |
| | RAPIDLY inflate the BP cuff – 60 mm Hg above systolic BL not less than 200 |

If occlusion is incomplete, increase pressure by 50 mm Hg, up to 300 mm Hg

| | Mark start time: | | |
|---|---|---|---|
| | Occlusion start time::_ Occlusion end time::_ | <u> </u> | |
| | <ul> <li>Occlusion end time:</li></ul> | <u> </u> | |
| | Occlusion Release | | |
| | After exactly 5 minutes | | |
| | Rapidly release | | |
| | Lower gain of occluded arm to fit scre | een | |
| Phase | e 3—Test End | | |
| | Post Occlusion: change gain back | | |
| | Record 5 minutes post occlusion (no | less than 5 minutes) | |
| | Inform patient that you are about to e | | |
| | Click "Stop" | | |
| | Probes will deflate automatically, rem<br>Remove cuff | ove used probes, tape a | and discard |
| Blood<br>end of | pressure #3:/ (mm Hg)<br>f test: °F | HR (beats/min | n) Room Temp @ |
| Result | t (RHI): | Number of Leaks: | |
| Comm | nents: | | |
| PAT p | performed by: (please print) | | |
| Signa | iture: | | nte: / / |


























## 21.7 Invasive Coronary Reactivity Testing – Screening and Month 6

Screening (if needed) and Month 6 CRT will be performed

### Pre-Angiogram CRT Instructions

- 1. Please fast before your appointment.
  - Nothing to eat or drink for 12 hours prior to your appointment (except you may drink water.
  - No caffeine 24 hours prior to your appointment whenever possible (i.e. tea, coffee, chocolate, soda, Anacin/Excedrin).
- 2. Please discontinue your use of:
  - Nicotine 4 hrs prior to your appointment
  - Long-acting nitrates, short-acting calcium channel blockers, alpha blockers and beta blockers, ACE/ARB inhibitors, Renin and Aldosterone Inhibitors for 24 hours prior to your testing whenever possible
  - Long-acting calcium channel blockers for 48 hours prior to your testing.
  - Sublingual nitroglycerin for 4 hours prior to your testing.
  - . Bring your medications with you so that you can take them after the procedure.

### Cath Lab requirements

- 1. Catheter size (e.g. 6 Fr) must be indicated
- Flags on all cine runs
- Obtain baseline angio (contrast injection) with the flow-wire in place



 12-lead EKG recording during infusions to evaluate for ST/T changes and documentation of chest pain

# **Diagnostic Coronary Angiography**

- 1. Insert 7F sheath in the femoral artery.
- Diagnostic left and right coronary angiography
- Measure LVEDP using pigtail catheter

## Coronary Reactivity Testing

- Once equipment is set up and flow wire is in position start the Volcano Machine timer (Press Baseline 2 times to start timer).
- Set Volcano Machine to either "Split screen" or "full screen" view according to local preference.
- Investigator to choose vessel for testing. Make sure the vessels are not overlapping, ECG leads are not obstructing view and vessel is adequately filled when obtaining cine images.
- Take baseline Angiogram marked as "Baseline"
- Record baseline Cine View this includes documentation of angles and cath size being used
- 5. Set Doppler in CFR mode
  - a. Record baseline blood pressure/heart rate
  - b. Press "Baseline" on Volcano Machine/Record baseline APV
  - d. Record infusion time
  - e. Flush
  - f. wait 5 seconds
  - g. Press "PEAK" on Volcano Machine
  - h. Wait for peak CFR to appear.
  - Record peak blood pressure/heart rate/ Peak APV/CFR
  - Press print.
  - a. Record baseline blood pressure/heart rate
  - b. Press "Baseline" on Volcano Machine/Record baseline APV
  - d. Record infusion time
  - e Flush
  - f. wait 5 seconds
  - g. Press "PEAK" on Volcano Machine
  - h. Wait for peak CFR to appear.
  - Record peak blood pressure/heart rate/ Peak APV/CFR
  - Press print.

- a. Record baseline blood pressure/heart rate
- b. Press "Baseline" on Volcano Machine/Record baseline APV
- d. Record infusion time
- e. Flush
- f. wait 5 seconds
- g. Press "PEAK" on Volcano Machine
- h. Wait for peak CFR to appear
- Record Peak blood pressure/heart rate/ Peak APV/CFR
- Press print.
- NOTE 1: May repeat any of the doses at the investigator's discretion
- NOTE 2: The highest CFR value from all the measurements will be used to qualify the subject for eligibility

- To program machine, press "System On".
- 3. "New Patient" press Yes
- 4. "Telemetry" or "Adult ICU" press Yes
- 5. Machine will auto-detect syringe. Select syringe and press "Confirm"
- Select "Rate" and enter 60 (mL/hr)
- 7. Select "VTBI" and enter 2.4 (mL)
- Press "Options" select "Anesthesia Mode" select "Enable"
- Press "Start" to start infusion
- 10. When infusion is complete, pump will beep. Press "Silence"

## reconnect tubing

- 12. Press "Channel select" on pump
- 13. IV machine will prompt again for syringe, select and "Confirm"
- 14. Press "Restore"
- 15. Press "Start" to begin second infusion

NOTE: Infuse into the catheter dead space 3.5 cc (infusion catheter space: 3 cc; infusion stopcock: 0.5 cc)

- 1. Set Volcano on "Trend Mode"
- Make sure pump is attached to the IV pole and hand sterile tubing to angiographer
- Select the syringe size (usually only choice of BD 10 cc syringe) and press "Confirm"
- Enter infusion rate "60" cc/hr (this will distribute the dose over 3 minutes) and VTBI "2.4" cc (this will deliver 2 cc intracoronary)
  - a. Record baseline blood pressure/heart rate
  - b. Press Baseline on Volcano Machine/Record baseline APV
  - c. Start timer for 3 min/record time on Volcano Machine
  - e. Image Cine Marker during infusion- "ACH low" or "10-6"
  - f. At 2:50 minutes press PEAK on Volcano Machine
  - g. Wait for peak CFR to appear
  - h. Record Peak blood pressure/heart rate/ Peak APV/CFR
  - i. Press print

in the infusion catheter prior to cine

k. Take cine image

- 10. Press "Channel Select" again once loaded, and "Confirm" syringe (20 cc syringe)
- 11. Press "Restore" for prior settings and "Start" when ready to infuse
  - a. Record baseline blood pressure/heart rate
  - b. Press Baseline on Volcano Machine/Record baseline APV
  - Start timer for 3 min/record time on Volcano Machine

- f. At 2:50 minutes press PEAK on Volcano Machine
- g. Wait for peak CFR to appear
- h. Record Peak blood pressure/heart rate/ Peak APV/CFR
- Press print
- Angiographer will clear 3 cc of high-dose acetylcholine prior to cine
- k. Take cine image
- Set Volcano to "Split screen"
- Place Cine Marker- "NTG"
- Record baseline blood pressure/heart rate
- Press Baseline on Volcano Machine/Record baseline APV
- 6. Flush
- 7. At 30 seconds press "PEAK" on Volcano Machine
- 8. Wait for peak CFR to appear.
- Record peak blood pressure/heart rate/Peak APV/CFR
- 10. Press print
- 11. Take Cine Image immediately after Peak APV/CFR is recorded

## 21.8 Cell Delivery Protocol

# Pre-Angiogram Cell Delivery Subject Instructions

- Please fast before your appointment.
  - Nothing to eat or drink for 12 hours prior to your appointment (except you may drink water).
- Please discontinue your use of:
  - Nicotine 4 hrs prior to your appointment
  - Bring your medications with you so that you can take them after the procedure.

#### Cath Lab requirements

- 1. Catheter size (e.g. 6 Fr) must be indicated
- Obtain LAD baseline angio (contrast injection)
- Infusion catheter will be the LAD seating catheter

### **Cell Delivery**

The general procedure for administration of CLBS16 is provided below. Please refer to the investigational product manual for this protocol for specific details.



#### 22. SIGNIFICANT CHANGES FROM PROTOCOL VERSION 6



### 23. REFERENCES

- Garg R, Rao AD, Baimas-George M, Hurwitz S, Foster C, Shah RV, Jerosch-Herold M, Kwong RY, Di Carli MF, and Adler GK, Mineralocorticoid receptor blockade improves coronary microvascular function in individuals with type 2 diabetes. Diabetes, 2015. 64(1): p. 236-242.
- Pauly DF, Johnson BD, Anderson RD, Handberg EM, Smith KM, Cooper-DeHoff RM, Sopko G, Sharaf BM, Kelsey SF, Merz CN, and Pepine CJ, In women with symptoms of cardiac ischemia, nonobstructive coronary arteries, and microvascular dysfunction, angiotensin-converting enzyme inhibition is associated with improved microvascular function: A double-blind randomized study from the National Heart, Lung and Blood Institute Women's Ischemia Syndrome Evaluation (WISE). Am Heart J, 2011. 162(4): p. 678-684.
- Pepine CJ, Ferdinand KC, Shaw LJ, Light-McGroary KA, Shah RU, Gulati M, Duvernoy C, Walsh MN, Bairey Merz CN, and Committee ACiW, Emergence of Nonobstructive Coronary Artery Disease: A Woman's Problem and Need for Change in Definition on Angiography. J Am Coll Cardiol, 2015. 66(17): p. 1918-1933.
- Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG, and Douglas PS, Low diagnostic yield of elective coronary angiography. N Engl J Med, 2010. 362(10): p. 886-895.
- Radico F, Cicchitti V, Zimarino M, and De Caterina R, Angina pectoris and myocardial ischemia in the absence of obstructive coronary artery disease: practical considerations for diagnostic tests. JACC Cardiovasc Interv, 2014. 7(5): p. 453-463.
- Jespersen L, Hvelplund A, Abildstrom SZ, Pedersen F, Galatius S, Madsen JK, Jorgensen E, Kelbaek H, and Prescott E, Stable angina pectoris with no obstructive coronary artery disease is associated with increased risks of major adverse cardiovascular events. Eur Heart J, 2012. 33(6): p. 734-744.
- Jespersen L, Abildstrom SZ, Hvelplund A, Galatius S, Madsen JK, Pedersen F, Hojberg S, and Prescott E, Symptoms of angina pectoris increase the probability of disability pension and premature exit from the workforce even in the absence of obstructive coronary artery disease. Eur Heart J, 2013. 34(42): p. 3294-3303.
- Shaw LJ, Merz CN, Pepine CJ, Reis SE, Bittner V, Kip KE, Kelsey SF, Olson M, Johnson BD, Mankad S, Sharaf BL, Rogers WJ, Pohost GM, Sopko G, and Women's Ischemia Syndrome Evaluation I, The economic burden of angina in women with suspected ischemic heart disease: results from the National Institutes of Health--National Heart, Lung, and Blood Institute--sponsored Women's Ischemia Syndrome Evaluation. Circulation, 2006. 114(9): p. 894-904.
- Camici PG and Crea F, Coronary microvascular dysfunction. N Engl J Med, 2007. 356(8): p. 830-840.
- Phan A, Shufelt C, and Merz CN, Persistent chest pain and no obstructive coronary artery disease. JAMA, 2009. 301(14): p. 1468-1474.
- Murthy VL, Naya M, Taqueti VR, Foster CR, Gaber M, Hainer J, Dorbala S, Blankstein R, Rimoldi O, Camici PG, and Di Carli MF, Effects of sex on coronary

- microvascular dysfunction and cardiac outcomes. Circulation, 2014. 129(24): p. 2518-2527.
- Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR, Jr., and Lerman A, Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation, 2000. 101(9): p. 948-954.
- Sara JD, Widmer RJ, Matsuzawa Y, Lennon RJ, Lerman LO, and Lerman A, Prevalence of Coronary Microvascular Dysfunction Among Patients With Chest Pain and Nonobstructive Coronary Artery Disease. JACC Cardiovasc Interv, 2015. 8(11): p. 1445-1453.
- Heistad DD, Armstrong ML, Marcus ML, Piegors DJ, and Mark AL, Augmented responses to vasoconstrictor stimuli in hypercholesterolemic and atherosclerotic monkeys. Circ Res, 1984. 54(6): p. 711-718.
- Sambuceti G, Marzullo P, Giorgetti A, Neglia D, Marzilli M, Salvadori P, L'Abbate A, and Parodi O, Global alteration in perfusion response to increasing oxygen consumption in patients with single-vessel coronary artery disease. Circulation, 1994. 90(4): p. 1696-1705.
- Sellke FW, Friedman M, Dai HB, Shafique T, Schoen FJ, Weintraub RM, and Johnson RG, Mechanisms causing coronary microvascular dysfunction following crystalloid cardioplegia and reperfusion. Cardiovasc Res, 1993. 27(11): p. 1925-1932.
- Gimelli A, Schneider-Eicke J, Neglia D, Sambuceti G, Giorgetti A, Bigalli G, Parodi G, Pedrinelli R, and Parodi O, Homogeneously reduced versus regionally impaired myocardial blood flow in hypertensive patients: two different patterns of myocardial perfusion associated with degree of hypertrophy. J Am Coll Cardiol, 1998. 31(2): p. 366-373.
- Pitkanen OP, Nuutila P, Raitakari OT, Ronnemaa T, Koskinen PJ, Iida H, Lehtimaki TJ, Laine HK, Takala T, Viikari JS, and Knuuti J, Coronary flow reserve is reduced in young men with IDDM. Diabetes, 1998. 47(2): p. 248-254.
- Yokoyama I, Momomura S, Ohtake T, Yonekura K, Nishikawa J, Sasaki Y, and Omata M, Reduced myocardial flow reserve in non-insulin-dependent diabetes mellitus. J Am Coll Cardiol, 1997. 30(6): p. 1472-1477.
- Yokoyama I, Ohtake T, Momomura S, Nishikawa J, Sasaki Y, and Omata M, Reduced coronary flow reserve in hypercholesterolemic patients without overt coronary stenosis. Circulation, 1996. 94(12): p. 3232-3238.
- Wang L, Jerosch-Herold M, Jacobs DR, Jr., Shahar E, and Folsom AR, Coronary risk factors and myocardial perfusion in asymptomatic adults: the Multi-Ethnic Study of Atherosclerosis (MESA). J Am Coll Cardiol, 2006. 47(3): p. 565-572.
- Pepine CJ, Anderson RD, Sharaf BL, Reis SE, Smith KM, Handberg EM, Johnson BD, Sopko G, and Bairey Merz CN, Coronary microvascular reactivity to adenosine predicts adverse outcome in women evaluated for suspected ischemia results from the National Heart, Lung and Blood Institute WISE (Women's Ischemia Syndrome Evaluation) study. J Am Coll Cardiol, 2010. 55(25): p. 2825-2832.

- 23. Reis SE, Holubkov R, Lee JS, Sharaf B, Reichek N, Rogers WJ, Walsh EG, Fuisz AR, Kerensky R, Detre KM, Sopko G, and Pepine CJ, Coronary flow velocity response to adenosine characterizes coronary microvascular function in women with chest pain and no obstructive coronary disease. Results from the pilot phase of the Women's Ischemia Syndrome Evaluation (WISE) study. J Am Coll Cardiol, 1999. 33(6): p. 1469-1475.
- 24. Thomson LE, Wei J, Agarwal M, Haft-Baradaran A, Shufelt C, Mehta PK, Gill EB, Johnson BD, Kenkre T, Handberg EM, Li D, Sharif B, Berman DS, Petersen JW, Pepine CJ, and Bairey Merz CN, Cardiac magnetic resonance myocardial perfusion reserve index is reduced in women with coronary microvascular dysfunction. A National Heart, Lung, and Blood Institute-sponsored study from the Women's Ischemia Syndrome Evaluation. Circ Cardiovasc Imaging, 2015. 8(4).
- Agarwal M, Shufelt C, Mehta PK, Gill E, Berman DS, Li D, Sharif B, Li N, Bairey Merz CN, and Thomson LE, Cardiac risk factors and myocardial perfusion reserve in women with microvascular coronary dysfunction. Cardiovasc Diagn Ther, 2013. 3(3): p. 146-152.
- 26. Erbs S, Linke A, Schachinger V, Assmus B, Thiele H, Diederich KW, Hoffmann C, Dimmeler S, Tonn T, Hambrecht R, Zeiher AM, and Schuler G, Restoration of microvascular function in the infarct-related artery by intracoronary transplantation of bone marrow progenitor cells in patients with acute myocardial infarction: the Doppler Substudy of the Reinfusion of Enriched Progenitor Cells and Infarct Remodeling in Acute Myocardial Infarction (REPAIR-AMI) trial. Circulation, 2007. 116(4): p. 366-374.
- Schachinger V, Assmus B, Honold J, Lehmann R, Hofmann WK, Martin H, Dimmeler S, and Zeiher AM, Normalization of coronary blood flow in the infarctrelated artery after intracoronary progenitor cell therapy: intracoronary Doppler substudy of the TOPCARE-AMI trial. Clin Res Cardiol, 2006. 95(1): p. 13-22.
- Kawamoto A, Gwon HC, Iwaguro H, Yamaguchi JI, Uchida S, Masuda H, Silver M, Ma H, Kearney M, Isner JM, and Asahara T, Therapeutic potential of ex vivo expanded endothelial progenitor cells for myocardial ischemia. Circulation, 2001. 103(5): p. 634-637.
- Losordo DW, Henry TD, Davidson C, Sup Lee J, Costa MA, Bass T, Mendelsohn F, Fortuin FD, Pepine CJ, Traverse JH, Amrani D, Ewenstein BM, Riedel N, Story K, Barker K, Povsic TJ, Harrington RA, Schatz RA, and Investigators AC, Intramyocardial, autologous CD34+ cell therapy for refractory angina. Circ Res, 2011. 109(4): p. 428-436.
- Vrtovec B, Poglajen G, Lezaic L, Sever M, Domanovic D, Cernelc P, Socan A, Schrepfer S, Torre-Amione G, Haddad F, and Wu JC, Effects of intracoronary CD34+ stem cell transplantation in nonischemic dilated cardiomyopathy patients: 5-year follow-up. Circ Res, 2013. 112(1): p. 165-173.
- 31. Poglajen G, Sever M, Cukjati M, Cernelc P, Knezevic I, Zemljic G, Haddad F, Wu JC, and Vrtovec B, Effects of transendocardial CD34+ cell transplantation in

- patients with ischemic cardiomyopathy. Circ Cardiovasc Interv, 2014. 7(4): p. 552-559.
- Serruys PW, di Mario C, Piek J, Schroeder E, Vrints C, Probst P, de Bruyne B, Hanet C, Fleck E, Haude M, Verna E, Voudris V, Geschwind H, Emanuelsson H, Muhlberger V, Danzi G, Peels HO, Ford AJ, Jr., and Boersma E, Prognostic value of intracoronary flow velocity and diameter stenosis in assessing the shortand long-term outcomes of coronary balloon angioplasty: the DEBATE Study (Doppler Endpoints Balloon Angioplasty Trial Europe). Circulation, 1997. 96(10): p. 3369-3377.
- 33. Povsic TJ, Henry TD, Traverse JH, Fortuin FD, Schaer GL, Kereiakes DJ, Schatz RA, Zeiher AM, White CJ, Stewart DJ, Jolicoeur EM, Bass T, Henderson DA, Dignacco P, Gu Z, Al-Khalidi HR, Junge C, Nada A, Hunt AS, Losordo DW, and Investigators R, The RENEW Trial: Efficacy and Safety of Intramyocardial Autologous CD34(+) Cell Administration in Patients With Refractory Angina. JACC Cardiovasc Interv, 2016. 9(15): p. 1576-1585.
- Lezaic L, Socan A, Poglajen G, Peitl PK, Sever M, Cukjati M, Cernelc P, Wu JC, Haddad F, and Vrtovec B, Intracoronary transplantation of CD34(+) cells is associated with improved myocardial perfusion in patients with nonischemic dilated cardiomyopathy. J Card Fail, 2015. 21(2): p. 145-152.
- 35. Wang S, Cui J, Peng W, and Lu M, Intracoronary autologous CD34+ stem cell therapy for intractable angina. Cardiology, 2010. 117(2): p. 140-147.
- Musialek P, Tekieli L, Kostkiewicz M, Majka M, Szot W, Walter Z, Zebzda A, Pieniazek P, Kadzielski A, Banys RP, Olszowska M, Pasowicz M, Zmudka K, and Tracz W, Randomized transcoronary delivery of CD34(+) cells with perfusion versus stop-flow method in patients with recent myocardial infarction: Early cardiac retention of (9)(9)(m)Tc-labeled cells activity. J Nucl Cardiol, 2011. 18(1): p. 104-116.





Prognostic value of peripheral arterial tonometry in patients with coronary artery disease and a high cardiovascular risk profile. J Atheroscler Thromb, 2014. 21(3): p. 230-238.

- 47. Wei J, Mehta PK, Johnson BD, Samuels B, Kar S, Anderson RD, Azarbal B, Petersen J, Sharaf B, Handberg E, Shufelt C, Kothawade K, Sopko G, Lerman A, Shaw L, Kelsey SF, Pepine CJ, and Merz CN, Safety of coronary reactivity testing in women with no obstructive coronary artery disease: results from the NHLBI-sponsored WISE (Women's Ischemia Syndrome Evaluation) study. JACC Cardiovasc Interv, 2012. 5(6): p. 646-653.
- 48. Campeau L, Grading of angina pectoris (letter). Circulation, 1976. 54: p. 522-523.
- Campeau L, The Canadian Cardiovascular Society grading of angina pectoris revisited 30 years later. Can J Cardiol, 2002. 18(4): p. 371-379.

#### INVESTIGATOR ACKNOWLEDGEMENT

An Open-Label Exploratory Clinical Study to Evaluate the Safety and Potential Bioactivity of CLBS16 in Patients with Coronary Microvascular Dysfunction and Without Obstructive Coronary Artery Disease

PROTOCOL NUMBER: CLBS16-P01
ClinicalTrials.gov Identifier: NCT03508609
Version Number: 7

Version Date: 26 August 2019

By signing below, the investigator acknowledges that he/she has read and understands this protocol and provides assurance that this study will be conducted according to all requirements as defined in this protocol, clinical study agreement, ICH GCP guidelines, and all applicable regulatory requirements.

| Investigator Signature | Date | - |
|--------------------------------------|------|---|
| Print Name and Title of Investigator | | |